CLINICAL TRIAL: NCT07105644
Title: Observational Study of Sacral Nerve Function After Sacral Tumor Resection
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 25SL016
Record Dates: First submitted 2025-07-08; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-06

CONDITIONS: Sacral Tumors
Keywords: sacral nerve function; motor functions; bowel functions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sacral Tumor Resection Post-Surgery Cohort: This cohort consists of patients diagnosed with sacral tumors (either primary or metastatic) who have undergone sacral tumor resection surgery. The study focuses on evaluating the post-surgical impact on motor functions, bowel functions, bladder functions, and overall quality of life. Patients in this cohort will be monitored for functional outcomes at various time points post-surgery (2 weeks, 3 months, 6 months, and 12 months). The study also includes a comprehensive assessment of neurological function based on sacral nerve preservation during surgery, including neural root sacrifice and the level of sacral resection performed.

SUMMARY:
The goal of this observational study is to evaluate the long-term effects of sacral tumor resection on sacral nerve function in patients with primary sacral tumors, including chordomas and chondrosarcomas. The study will primarily focus on understanding how the level of sacral resection impacts postoperative motor, bowel, bladder, and sexual functions. The main questions it aims to answer are:

How does the level of sacral resection influence bowel and bladder function at 12 months post-surgery? What is the role of preserving the sacral nerve root in maintaining motor function and sexual function? Participants will include patients who have undergone sacral tumor resection and will be followed for 12 months post-surgery. They will provide data on their bowel, bladder, and motor functions, as well as sexual function, through clinical evaluations and standardized questionnaires.

Participants will:

Complete surveys on bowel, bladder, and motor function at baseline and at 3, 6, and 12 months after surgery Undergo clinical assessments, including anorectal manometry, post-void residual urine volume measurements, and sensory evaluations Be evaluated for changes in sexual function using standardized surveys like IIEF (for males) and FSFI (for females)

DETAILED DESCRIPTION:
This observational study is designed to assess the long-term impact of sacral tumor resection on sacral nerve function in patients diagnosed with primary sacral tumors, such as chordomas and chondrosarcomas. The objective is to determine the relationship between the level of sacral resection and the preservation of bowel, bladder, motor, and sexual functions post-surgery. The study will track functional recovery over 12 months, focusing on how different resection levels affect these outcomes.

The study will include patients who undergo sacral tumor resection with varying degrees of nerve root sacrifice. Participants will be categorized based on the extent of resection: those who undergo a low sacrectomy and those who undergo a high sacrectomy.

The primary research questions are:

How does the level of sacral resection (low, middle, high, or total) impact functional outcomes such as bowel, bladder, motor, and sexual function at 12 months post-surgery?

How does the preservation of the sacral nerve root affect functional recovery compared to the sacrifice of this nerve root?

To address these questions, participants will complete a series of standardized questionnaires at baseline, 3 months, 6 months, and 12 months after surgery to assess:

Bowel Function: Evaluated using anorectal manometry and the Cleveland Constipation Score and Wexner Incontinence Score.

Bladder Function: Assessed through ICIQ-SF (bladder function), Saito grading, and urodynamic tests (e.g., maximum urinary flow, post-void residual urine).

Motor Function: Evaluated through Frankel scores and mobility assessments.

Sexual Function: Measured using the IIEF for males and the FSFI for females.

This study will provide important data on the functional outcomes of sacral tumor resection, helping to guide clinical decisions on surgical techniques and post-surgical management to optimize patient recovery and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Age between 12 and 80 years Confirmed diagnosis of sacral tumor (either a primary bone tumor or a metastatic tumor from another solid malignancy) Able to understand the study requirements and provide written informed consent

Exclusion Criteria:

Poor general condition rendering the patient unable to tolerate surgery History of diseases or surgeries affecting bowel or bladder function Missing intraoperative data regarding sacral resection level or nerve root sacrifice Pregnant or currently breastfeeding Missing critical follow-up data or lost to follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients aged 12 to 80 years diagnosed with sacral tumors (either primary bone tumors or metastases from other solid tumors) who are scheduled for surgical resection at Shanghai Changzheng Hospital. All participants must meet inclusion criteria and provide informed consent. The study will assess postoperative motor, bowel, and bladder function, pain, quality of life, and complications. Patients unable to tolerate surgery or with pre-existing bowel/bladder dysfunction will be excluded. A total of 400 patients will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Bladder Function Score at 12 Months Post-Surgery | 12 months post-surgery: Bladder function will be assessed during a comprehensive follow-up visit at 12 months after the surgery.
  The primary outcome measure will assess bladder function 12 months after sacral tumor resection surgery. Based on the Biagini et al. method and supported by literature such as Huang et al the bladder function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to micturate and has limited continence at varying times and quantities of urine and/or has increasing postmicturition vesical residual and/or urinary loss in conditions of stress
  2. Does not feel stimulus to micturate and/or is completely incontinent

SECONDARY OUTCOMES:
Rectal Function Score at 12 Months Post-Surgery | 12 months post-surgery: Rectal function will be assessed during a follow-up visit at 12 months after the surgery.
  The secondary outcome measure will assess rectal function 12 months after sacral tumor resection surgery. Based on the Biagini et al. method and supported by literature such as Huang et al the Rectal function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to defecate and is incontinent when feces are soft or under stress
  2. Does not feel stimulus to defecate and/or is completely incontinent

OTHER OUTCOMES:
Pre-Surgical Baseline Information-Age | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  Patient age at the time of surgery, recorded in years as a continuous variable.
Pre-Surgical Baseline Information-Gender | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  Patient sex as recorded in the medical record (male or female).
Pre-Surgical Baseline Information-Time from Treatment Initiation to First Diagnosis | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  The duration, in months, between the initiation of any relevant prior treatment (e.g., symptomatic management, imaging, or biopsy) and the date of histopathological diagnosis of sacral tumor
Pre-Surgical Baseline Information-Body Mass Index (BMI) | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  Calculated as weight in kilograms divided by height in meters squared (kg/m²), recorded as a continuous variable.
Pre-Surgical Baseline Information-Pre-Surgical Treatment History | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  Documentation of any tumor-related treatments received prior to surgery, including radiotherapy, chemotherapy, embolization, or prior surgical interventions.
Pre-Surgical Baseline Information-ECOG Performance Status | 2 days before surgery: The pre-surgical baseline information will be collected during the patient's preoperative assessment, which will occur 2 days before the surgery.
  Patient performance status at the time of enrollment, scored using the Eastern Cooperative Oncology Group (ECOG) scale (range: 0 to 5), where higher scores indicate worse functional impairment.
Pre-Rectal Function Score | 2 days before surgery: Bowel function will be assessed during the preoperative assessment conducted 2 days before the surgery.
  The secondary outcome measure will assess rectal function 12 months after sacral tumor resection surgery. Based on the Biagini et al. method and supported by literature such as Huang et al the Bowel function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to defecate and is incontinent when feces are soft or under stress
  2. Does not feel stimulus to defecate and/or is completely incontinent
Pre-Bladder Function Score | 2 days before surgery: Urinary function will be assessed during the preoperative assessment conducted 2 days before the surgery.
  Based on the Biagini et al. method and supported by literature such as Huang et al the bladder function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to micturate and has limited continence at varying times and quantities of urine and/or has increasing postmicturition vesical residual and/or urinary loss in conditions of stress
  2. Does not feel stimulus to micturate and/or is completely incontinent
Pre-Surgical Pain Assessment (VAS Score) | 2 days before surgery: Pain will be assessed using the VAS during the preoperative assessment conducted 2 days before the surgery.
  This outcome measure will assess pain levels prior to surgery using the Visual Analog Scale (VAS). The VAS is a widely used tool for measuring the intensity of pain, with patients indicating their level of pain on a scale from 0 (no pain) to 10 (worst possible pain). This pre-surgical pain assessment will provide a baseline for understanding the patient's pain levels, which will be compared to post-surgical pain levels to assess recovery and the effectiveness of post-operative pain management.
Intra-Surgical Data Collection-Surgical Time | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Total duration of the surgical procedure, measured in minutes from initial incision to closure.
Intra-Surgical Data Collection-Blood Loss | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Estimated total volume of intraoperative blood loss, recorded in milliliters (mL).
Intra-Surgical Data Collection-Surgical Approach | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  The operative corridor used to access the tumor, classified as anterior, posterior, or combined anterior-posterior approach.
Intra-Surgical Data Collection-Implantation of Internal Fixation | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Whether spinal or pelvic instrumentation (e.g., screws, rods) was implanted during surgery (yes or no).
Intra-Surgical Data Collection-Highest Sacral Resection Level | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  The most cephalad sacral vertebral level at which osteotomy was performed, based on intraoperative and radiographic records (e.g., S1, S2, S3, etc.).
Intra-Surgical Data Collection-Nerve Root Ligation | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  The number and laterality (unilateral/bilateral) of sacral nerve roots ligated or sacrificed during tumor resection, documented per operative report.
Intra-Surgical Data Collection-Tumor Resection Technique | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Type of surgical excision performed, categorized as en bloc resection or piecemeal resection.
Intra-Surgical Data Collection-Intraoperative Bowel Involvement | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Whether the tumor showed direct involvement or adherence to the bowel, as identified during surgery (yes or no).
Intra-Surgical Data Collection-Vascular Adhesions | During Surgery: These data points will be collected in real-time during the surgery and documented by the surgical team.
  Presence of tumor adhesion to major pelvic vessels observed intraoperatively, as judged by the operating surgeon (yes or no).
Post-Surgical Rectal Function Score | 3 months post-surgery6 months post-surgery
  The secondary outcome measure will assess rectal function 12 months after sacral tumor resection surgery. Based on the Biagini et al. method and supported by literature such as Huang et al the Bowel function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to defecate and is incontinent when feces are soft or under stress
  2. Does not feel stimulus to defecate and/or is completely incontinent
Post-Surgical bladder Function Score | 3 months post-surgery6 months post-surgery
  Based on the Biagini et al. method and supported by literature such as Huang et al the bladder function scoring system commonly used in sacrectomy outcome studies includes the following components:
  0-Normal
  1. Feels stimulus to micturate and has limited continence at varying times and quantities of urine and/or has increasing postmicturition vesical residual and/or urinary loss in conditions of stress
  2. Does not feel stimulus to micturate and/or is completely incontinent
Post-Surgical Pain Assessment (VAS Score) | 2 weeks post-surgery3 months post-surgery6 months post-surgery12 months post-surgery
  Postoperative pain intensity is assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Patients are asked to report their daily worst pain. All patients receive standardized NSAID treatment. If additional opioid analgesics are used, the VAS score prior to opioid administration and the dose of opioid used are recorded. Higher scores indicate more severe pain
Post-Surgical Quality of Life (QLQ-C30) | 2 weeks post-surgery3 months post-surgery6 months post-surgery12 months post-surgery
  Health-related quality of life is evaluated using the EORTC QLQ-C30 questionnaire, a validated 30-item instrument developed by the European Organisation for Research and Treatment of Cancer. It includes five functional domains, three symptom domains, a global health status score, and additional symptom items. Scores range from 0 to 100. For functional and global health domains, higher scores indicate better function; for symptom domains, higher scores indicate more severe symptoms.
Post-Surgical Disease Control-Progression-Free Survival (PFS) | Post-Surgery: Disease control and adjuvant treatment will be assessed at 3 months, 6 months, and 12 months post-surgery, with regular follow-up to monitor tumor status and treatment effects.
  Defined as the time interval from the date of surgery to the date of radiologically or clinically confirmed tumor progression or recurrence, as assessed by postoperative MRI and/or symptom evaluation. Patients without progression at the time of last follow-up will be censored.
Post-Surgical Disease Control-Progression-Overall Survival (OS) | Post-Surgery: Disease control and adjuvant treatment will be assessed at 3 months, 6 months, and 12 months post-surgery, with regular follow-up to monitor tumor status and treatment effects.
  Defined as the time from surgery to death from any cause. Patients alive at the time of last follow-up will be censored.
Adjuvant Treatment | Post-Surgery: Disease control and adjuvant treatment will be assessed at 3 months, 6 months, and 12 months post-surgery, with regular follow-up to monitor tumor status and treatment effects.
  Documentation of any postoperative oncologic therapy, including radiotherapy, chemotherapy, targeted therapy, or immunotherapy. Treatment modality, agent used, and combination strategy (if any) are recorded.
Treatment Duration | Post-Surgery: Disease control and adjuvant treatment will be assessed at 3 months, 6 months, and 12 months post-surgery, with regular follow-up to monitor tumor status and treatment effects.
  Duration of each adjuvant therapy regimen (in days), recorded from initiation to completion or discontinuation. Reasons for discontinuation, if applicable (e.g., toxicity, progression), are documented.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Doctor, Study Director — Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) may not be shared in this study due to the following reasons:
  Confidentiality and Privacy Concerns: The study involves sensitive medical information related to patients' personal health, and sharing this data could compromise participant confidentiality. All data collected will be securely stored and accessed only by authorized personnel, in line with ethical standards and legal requirements.
  Ethical Considerations: Participants have provided informed consent for their data to be used solely for the purposes of this specific study. Sharing IPD outside of this scope might not align with the consent provided by participants.
  Regulatory and Institutional Policies: Institutional or regulatory policies may restrict the sharing of IPD to protect patient privacy and adhere to local laws, such as those related to data protection (e.g., GDPR in Europe or HIPAA in the United States).

REFERENCES:
- [Background] Phukan R, Herzog T, Boland PJ, Healey J, Rose P, Sim FH, Yazsemski M, Hess K, Osler P, DeLaney TF, Chen YL, Hornicek F, Schwab J. How Does the Level of Sacral Resection for Primary Malignant Bone Tumors Affect Physical and Mental Health, Pain, Mobility, Incontinence, and Sexual Function? Clin Orthop Relat Res. 2016 Mar;474(3):687-96. doi: 10.1007/s11999-015-4361-3. PMID 26013155
- [Background] Moran D, Zadnik PL, Taylor T, Groves ML, Yurter A, Wolinsky JP, Witham TF, Bydon A, Gokaslan ZL, Sciubba DM. Maintenance of bowel, bladder, and motor functions after sacrectomy. Spine J. 2015 Feb 1;15(2):222-9. doi: 10.1016/j.spinee.2014.08.445. Epub 2014 Sep 6. PMID 25195977

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/44/NCT07105644/Prot_SAP_ICF_000.pdf